CLINICAL TRIAL: NCT04721860
Title: Optimizing Training in Severe Post-Stroke Walking Impairment
Acronym: BLT2b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Oluwole Awosika, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0784
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Chronic Stroke; Walking, Difficulty; Gait, Hemiplegic
Keywords: Gait; Balance; Non-body weight supported treadmill training; Backward locomotion treadmill training; Forward locomotion treadmill training; Walking Rehabilitation; Walking Recovery
MeSH Terms: conditions — Stroke; Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Stratified Randomization
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Backward Locomotion Treadmill Training (BLTT) (Experimental): Participants train on a reverse treadmill (no bodyweight support), three times per week x 4 weeks.
  Interventions: Behavioral: Backward Locomotion Treadmill Training (BLTT)
- Forward Locomotion Treadmill Training (FLTT) (Sham Comparator): Participants train on a treadmill (no bodyweight support), three times per week x 4 weeks.
  Interventions: Behavioral: Forward Locomotion Treadmill Training (FLTT)

INTERVENTIONS:
Behavioral: Backward Locomotion Treadmill Training (BLTT) — 12-training sessions of reverse treadmill training (no bodyweight support) over four weeks.
  Arms: Backward Locomotion Treadmill Training (BLTT)
Behavioral: Forward Locomotion Treadmill Training (FLTT) — 12-training sessions of forward treadmill training (no bodyweight support) over tfour weeks.
  Arms: Forward Locomotion Treadmill Training (FLTT)

SUMMARY:
Difficulty walking is common after a stroke. Although physical rehabilitation helps a little with the improvement of walking ability, recovery is usually incomplete. The purpose of this study is to explore how two different treadmill training approaches influence walking speed, symmetry, and balance in people with chronic severe stroke-related walking impairment. The two approaches involve either forward or backwards treadmill training. This study will look at changes in walking performance and balance, before and after training. This study may lead to more efficient methods for improving walking performance and balance after stroke.

DETAILED DESCRIPTION:
Severe walking impairment after stroke is defined as the inability to walk faster than 0.4 meters per second and impacts nearly twenty-five percent of chronic stroke survivors. Walking speed is a key determiner of community independence, and stroke survivors classified as "severe" are more often symptomatically home-bound with limited mobility and are at higher risk of falls, fractures, and rehospitalizations. A recent study by the investigators suggests that backward locomotion treadmill training (BLTT) may be a promising rehabilitative approach in stroke survivors with severe walking impairment; however, the effect of training duration on behavioral outcomes is unknown.

The objective of this study is to obtain critical pilot data on the effects of extended BLTT on walking speed, symmetry, and balance (static and dynamic), in chronic stroke survivors with baseline severe walking impairment, relative to forward treadmill training controls (FLTT).

Aim 1. Determine the training-related effects of extended BLTT on overground walking speed (primary outcome) in survivors with severe walking impairment. To achieve this aim, we will compare the Pre-Post change in walking speed [10- meter walk test (10MWT)] between groups. The working hypothesis is that extended BLTT will increase walking speed to a clinically meaningful level (≥0.16m/s), compared to the control group (FLTT).

Aim 2. Determine the effects of extended BLTT on walking symmetry and balance. The Zeno Walkway Gait Analysis software will capture Pre-Post changes in temporal gait symmetry index during the 10-MWT. Working hypothesis 2a: BLTT will be associated with a favorable improvement in the temporal symmetry index score. Proprioception and spinovestibular function will be measured with the modified Sensorineural Integration Test (mSIT), and dynamic balance will be assessed with the completion time on the instrumented Timed Up & Go (i- TUG). Working hypothesis 2b and c: BLTT will be associated with a favorable improvement Pre-Post mSIT(a) and completion time on the i-TUG (b).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Walking speed less than or equal to 0.4 meters/second
* Ability to maintain greater than or equal to 0.3mph speed for 6-minute interval on the treadmill
* Able to walk independently (cane and hemi-walker acceptable)
* Ambulate >10 meters over ground with the Free Step Harness System (as a safety precaution)
* Discharged from formal rehabilitation

Exclusion Criteria:

* Unstable cardiac status which would preclude participation in a moderate-intensity exercise program.
* Significant language barrier which might prevent the participant from following instructions during training and testing.
* Adverse health condition that might affect walking capacity (severe arthritis, significant pulmonary disease significant ataxia, or severe hemi-neglect)
* Severe lower extremity spasticity (Ashworth >2)
* Depression (>10 on the Patient Health Questionnaire, if untreated).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in 10-Meter Walk (fast) | Pre-Baseline (Day of Randomization) to One Day Post-Training
  Two 10MWT trials (using a stop-watch) are averaged and documented in meters/second.

SECONDARY OUTCOMES:
10-Meter Walk Test (Fast- Retention) | One Day Post Training, One month Post Training, 3- Months Post Training
  Two 10MWT (fast) trials (using a stop-watch) are averaged and documented in meters/second.
10-Meter Walk (Comfortable) | Baseline (Day of Randomization), One Day Post-Training, One month Post Training, 3-Months Post Training
  Two 10MWT trials (using a stop-watch) are averaged and documented in meters/second.

OTHER OUTCOMES:
Temporal Symmetry Index | Temporal Symmetry Index
  %-limb support of the affected and unaffected leg, during the 10 MWT
Static Balance: Sway Index (SI) | Baseline (Day of Randomization), One Day Post-Training, One month Post Training, 3- Months Post Training
  The Biodex Modified Clinical Test of Sensory Interaction on Balance (mSIBT) is a well-validated balance system and has been used neurally intact and neurologically impaired individuals to objectively measure static balance. Compared to other measures of static balance, the mSIBT provides the added benefit of differentiating the contributions of the visual, proprioceptive and vestibular systems. Method: While on the platform (with safety harness), participants will stand with the hands at the side under 4 conditions (30 secs/condition):1) firm surface with the eyes open, 2) firm surface with the eyes closed, 3) compliant surface (foam) with the eyes open, 4) Compliant surface (foam) with the eyes closed. Three attempts will be average and documented as SI.
Dynamic Balance: Instrumented Timed Up & Go (i-TUG)- 3 Meter | Baseline, One Day Post-Training, One month Post Training, 3- Months Post Training
  Participants will be instructed to sit with the back against the chair (seat height 46cm, arm height 67cm) and on the word "go," stand up, walk at a comfortable speed past the 3-m mark, turn around, walk back, and sit down in the chair. Two trials are averaged and documented in seconds.
Dynamic Balance: Instrumented Timed Up & Go (i-TUG)- 7 Meter | Baseline, One Day Post-Training, One month Post Training, 3- Months Post Training
  Participants will be instructed to sit with the back against the chair (seat height 46cm, arm height 67cm) and on the word "go," stand up, walk at a comfortable speed past the 7-m mark, turn around, walk back, and sit down in the chair. Two trials are averaged and documented in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No